CLINICAL TRIAL: NCT02284841
Title: Effect of Hilotherm Therapy on Post-operative Pain and Swelling Following Surgical Lower Third Molar Removal
Brief Title: Effect of Hilotherm Therapy on Post-operative Pain and Swelling Following Surgical Wisdom Tooth Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Version 1
Record Dates: First submitted 2014-10-09; First posted 2014-11-06 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Molar, Third; Wisdom Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hilotherm cooling face mask (Experimental): Use of Hilotherm cooling face mask post-operatively following surgical wisdom tooth removal to evaluate the incidence of pain and swelling
  Interventions: Device: Hilotherm cooling face mask
- No Hilotherm (No Intervention): No intervention following surgical wisdom tooth removal (same patient), therefore the patient is their own control.

INTERVENTIONS:
Device: Hilotherm cooling face mask — Hilotherapy - use of an external cooling device; a facial mask through which water circulates at a controlled temperature, allowing continuous cooling of the face, and is thought to reduce post-operative swelling and pain.
  Arms: Hilotherm cooling face mask

SUMMARY:
This study evaluates the efficacy of Hilotherm therapy on the incidence of swelling and pain following the surgical removal of lower wisdom teeth. All participants will have two lower wisdom teeth removed, with the Hilotherm cooling face mask only applied to one side of the patients' face for 60 minutes post-operatively, thus the patient being their own control.

DETAILED DESCRIPTION:
How does Hilotherm therapy affect post-operative pain and swelling after surgical wisdom tooth removal?

Wisdom tooth removal is one of the most common minor oral surgical procedures. The most widely experienced post-operative complications include pain and swelling, and so any research into how these effects can be minimised is of utmost importance to improve the quality of care we can deliver to our patients.

Our research is investigating the efficacy of Hilotherm therapy, which uses pre-shaped plastic facial masks through which water circulates at a controlled temperature, to reduce the experience of post-operative pain and swelling.

The Hilotherm face mask will be placed immediately after the surgery, while the patient is in the recovery area and will be worn on ONE side of the face, this being randomised using a computer programme and decided at the time of surgery. It will be worn for one hour after wisdom tooth removal. We will then use 3D photography analysis of the patients face to assess the extent of swelling, their assessment of pain using a visual analogue scale, and their overall satisfaction with Hilotherm therapy. These measurements will be recorded at:

Day 0 - 60 minutes post-op after patient has worn Hilotherm cooling mask Day 3 Day 10 Day 24

The person analysing the 3D images will be blinded to the side of the intervention.

All patients undergoing wisdom tooth removal on both sides, of similar surgical difficulty, to be carried out under a General Anaesthetic of the Daycase Unit of One Hospital will be eligible. Both extractions will be carried out by the same surgeon. Participants who undergo complications during or after the procedure will be excluded from our study. Extractions which end up being too dissimilar will also be excluded, and patients unsuitable for use of the Hilotherm mask (for example allergies) will also not be considered. Any patients with immune system affecting diseases, and patients who suffer allergic reactions to pharmaceutical agents will also not be considered.

No other elements of treatment will be changed from normal protocol.

ELIGIBILITY:
Inclusion Criteria:

* any patients requiring bilateral lower third molars extracted of similar technical difficulty under general anaesthesia

Exclusion Criteria:

* any intra-operative complications
* any post-operative complications, including infection
* if the extractions end up being too dissimilar surgically
* any contra-indication to the Hilotherm mask
* patients with any immune system-affecting diseases
* patients with allergies to pharmaceutical drugs (eg. analgesics or antibiotics)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in post-operative swelling using 3D photography analysis | Day 0 (pre/60 min post op), Days 3, 10, 24.
  Extent of swelling on the side of wisdom tooth removal with the intervention compared with the side without the intervention
Change in pain intensity using visual analogue scale | Day 0 (60 min post-op), Days 3, 10, 24.
  Self-reported pain intensity using visual analogue scale at time intervals as above, comparing the side of wisdom tooth removal with intervention vs the side of wisdom tooth removal without intervention

SECONDARY OUTCOMES:
Patient satisfaction | Day 24
  Patient satisfaction questionnaire to ask them to assess and compare side with intervention versus side without intervention. Did they feel it made a big difference to their post-operative pain and swelling, and to the speed with which they felt they could return to normal life (eg work?)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Fan, PhD, FDSRSC, FRCSEd, FRCS OMFS, Principal Investigator — Kings College Hospital NHS Foundation Trust
Locations (1):
- Queen Marys Hospital, Kings College London NHS Foundation Trust, Sidcup, Kent, United Kingdom